CLINICAL TRIAL: NCT04957446
Title: A Clinical Histology Study Evaluating Biostimulatory Activity Longevity of Injectable Poly-L-Lactic Acid (Sculptra Aesthetic) for Facial Rejuvenation
Brief Title: Histology Study of Biostimulatory Activity of Injectable Poly-L-Lactic Acid (Sculptra Aesthetic)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sadick Research Group (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SRG-PLLA-02
Record Dates: First submitted 2021-06-22; First posted 2021-07-12 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-06

CONDITIONS: Nasolabial Fold; Facial Wrinkles
Keywords: nasolabial fold; facial wrinkles

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, double-blind single-center study. Subjects will be randomized to either Group 1 (Sculptra Aesthetic) or Group 2 Placebo (Saline solution).
Who Masked: Participant, Investigator
Masking Description: The investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Experimental): Subjects will receive 3 treatments of 1mL Poly-L-Lactic Acid (Sculptra Aesthetic)
  Interventions: Device: Sculptra Aesthetic
- Group 2 (Placebo Comparator): Subjects will receive 3 treatments of 1mL Saline solution.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Sculptra Aesthetic — Injectable implant containing microparticles of poly-L-lactic acid (PLLA)
  Arms: Group 1
Other: Placebo — Saline solution
  Arms: Group 2

SUMMARY:
The study device, Sculptra, is an injectable implant formulation of poly-L-lactic acid microbeads, approved by the FDA for treatment of facial fat loss (lipoatrophy of HIV disease). It is being used off-label by dermatologists to treat dermal defects, as a biologically active filler. Anecdotal evidence suggests that subjects' skin quality may improve as a result of poly-L-lactic acid injection. While this is not the primary goal of such treatments it is often seen and described as so called "Sculptra glow". Based upon the study doctor's experience global skin quality improvement includes radiance, smoothness and pigment uniformity as well as a decrease in skin redness and pore size. In this study we evaluate the existence of histopathological (microscopic examination of tissue) evidence that can explain the observed improvement of skin quality after poly-L-lactic acid injections. Specifically, we will use histopathologic techniques to investigate effects of Sculptra injections into human skin with regard to restoring skin health and epidermal thickness.

DETAILED DESCRIPTION:
Sculptra is a formulation of poly-L-lactic acid microbeads, approved by the FDA for treatment of facial fat loss (lipoatrophy of HIV disease). It is being used off-label by dermatologists to treat dermal defects, as a biologically active filler. Anecdotal evidence suggests that patients' skin quality may improve as a result of poly-L-lactic acid injection. While this is not the primary goal of such treatments it is often seen and described as so called "Sculptra glow".

Based upon the investigator's experience global skin quality improvement includes radiance, smoothness and pigment uniformity as well as a decrease of erythema index and pore size. In this study we evaluate the existence of histopathological evidence that can elucidate the observed improvement of skin quality after poly-L-lactic acid injections. Specifically we will use histopathologic techniques to investigate effects of Sculptra injections into human skin with regard to dermal remodeling and epidermal thickness.This is a randomized, controlled, double-blind single-center study. The treatment phase will consist of a baseline visit, visits at 4-week and 8-weeks during which eligible subjects will receive injections of 5 cc of poly-L-lactic acid (PLLA) for the treatment group or saline for the control group into both sides of the face.

Seven eligible subjects will receive injections of 5 cc of poly-L-lactic acid (PLLA) for the study treatment group and 3 subjects will receive saline for the control group into both sides of the face.

The biopsy portion of the study, a punch biopsy will be collected at 4 timepoints throughout the study: at baseline prior to study treatment one, 4 weeks post study treatment one, 48 hours post study treatment three, and 18 weeks post study treatment.

Participation is up to 28 weeks and will attend approximately 6 study visits. The subject participation period includes a screening period of up to 2 weeks, three injections at 4-week intervals, and a follow-up visit at 48 hours and 18 weeks after the last injection.

to evaluate the histological effect and the "duration" of repeated subcutaneous injections of poly-L-lactic acid (PLLA) on skin quality. As skin SRG-PLLA-02 quality improvement the histopathological analysis with assess expression of procollagen 1, CD31 (vessels), SMA (myofibroblasts), CD163 (macrophages), CD117 (mast cells), & Elastin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained including HIPAA authorization
* Healthy females an males between 30 and 65 years of age
* Subjects with Fitzpatrick photo skin types I-IV
* Subjects with shallow to deep nasolabial fold contour deficiencies or other facial wrinkles
* Subjects who agree not to have any procedures affecting facial wrinkles (e.g. filler, botulinum toxin, radiofrequency, laser, IPL, ultrasound) for the duration of the study
* Subjects who do agree not to have any other procedures affecting skin quality (microdermabrasion, peels, acne treatments, etc.) for the duration of the study
* Subjects who understand this study and are able to follow study instructions and are willing to attend the required study visits
* Subjects who agree to be photographed for research reasons and their identity may not be concealed in these photographs

Exclusion Criteria:

* Subjects who are pregnant, planning to become pregnant or breastfeeding. A urine pregnancy test will be done to rule out pregnancy
* Subjects of child-bearing potential who are not using an approved method of birth control (oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence). Females of non-childbearing potential are defined as post-menopausal (absence of menstrual bleeding for one year), hysterectomy or bilateral oophorectomy.
* Subjects who cannot understand or are not willing to comply with the requirements of the study
* Subjects who have a known allergy to poly-L-lactic acid, carboxymethylcellulose, non-pyrogenic mannitol or any anesthetic
* Subjects who have taken any NSAIDs (aspirin, ibuprofen, etc.) within 7 days before treatment
* Subjects who have taken acetaminophen 24 hours before treatment
* Subjects who have had fillers or botulinum toxin in the treatment area in the past 12 months
* Subjects who have had treatments with poly-L-lactic acid in the face at any time
* Subjects who have had any kind of facial dermabrasion, chemical peel, laser, or IPL treatment including superficial treatments for aesthetic reasons in the past 6 months or for the duration of the study
* Subjects who does not agree to avoid using tanning beds or intensive exposure to the sun 2 two weeks prior to each office visit.
* Subjects who have any dermatologic conditions including acne, rosacea, eczema, psoriasis, actinic keratosis, severe sun damage, infection or scars within the treatment area
* Subjects who have an active inflammatory process (skin eruptions such as cysts, pimples, rashes or hives) or infection within the treatment area
* Subjects who have any known cancer including skin cancers (basal cell carcinoma, squamous cell carcinoma and melanoma)
* Subjects who have had systemic corticosteroid therapy in the past 6 months or for the duration of the study
* Subjects with a known history of poor wound healing
* Subjects with a known history of keloids (excessive scarring)
* Subjects who are HIV positive
* Subjects who have an existing medical condition that the Investigator considers may put the subject at risk or compromise their participation in the study
* Subjects who have participated in another research study in the past 30 days
* Subjects who are currently involved in any injury litigation claims

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Histological effect | 12 weeks
  The primary outcome measure is defined as the degree of improvement in skin quality based on the expression of tissue markers measured by a blinded histopathologist.

SECONDARY OUTCOMES:
Skin Improvement | 18 weeks
  The secondary outcome measure is defined as the degree of improvement in skin quality measured by a blinded, trained evaluator using standardized pictures as well as live evaluations rated by a blinded investigator and the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sadick, M.D., Principal Investigator — Sadick Research Group
Locations (1):
- Michelle Malanga, New York, New York, United States